CLINICAL TRIAL: NCT03763812
Title: Explorative Study on the Inflammatory Response After Endovascular Aortic Aneurysm Repair and Endovascular Aneurysm Sealing.
Brief Title: Post Implant Syndrome After EVAR and EVAS (INSPIRE Study)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Nellix stent cannot be placed in patients yet.
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, Principal investigator, Rijnstate Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INSPIRE study
Record Dates: First submitted 2018-11-13; First posted 2018-12-04 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Abdominal Aortic Aneurysm; Inflammatory Response
Keywords: EVAR; EVAS; Post implant syndrome; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Masking Description: No masking since patients, doctor and researchers know if patients undergo EVAR or EVAS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Aneurysm Repair (EVAR) (Other): Patients scheduled for EVAR will be included and blood samples at 7 time points will be taken.
  Interventions: Procedure: Endovascular Aneurysm Repair (EVAR)
- Endovascular Aneurysm Sealing (EVAS) (Other): Patients scheduled for EVAS will be included and blood samples at 7 time points will be taken.
  Interventions: Procedure: Endovascular Aneurysm Sealing (EVAS)

INTERVENTIONS:
Procedure: Endovascular Aneurysm Repair (EVAR) — The following blood samples will be taken: WBC and circulating cytokines (TNF-α, Interleukin (IL)-1, 1RA, 6, 10, 18, CRP), Troponin T, HsTnT, NT-pro-BNP at these time points:
  * Before induction of anesthesia
  * At wound closure
  * 24 hours after surgery
  * 48 hours after surgery
  * 1 month after surgery
  * 6 months after surgery
  * 12 months after surgery
  Arms: Endovascular Aneurysm Repair (EVAR)
Procedure: Endovascular Aneurysm Sealing (EVAS) — The following blood samples will be taken: WBC and circulating cytokines (TNF-α, Interleukin (IL)-1, 1RA, 6, 10, 18, CRP), Troponin T, HsTnT, NT-pro-BNP at these time points:
  * Before induction of anesthesia
  * At wound closure
  * 24 hours after surgery
  * 48 hours after surgery
  * 1 month after surgery
  * 6 months after surgery
  * 12 months after surgery
  Arms: Endovascular Aneurysm Sealing (EVAS)

SUMMARY:
Retrospective data have shown that active sac management, as applied in EVAS, reduces the incidence of the post-implant syndrome. All-cause and cardiac mortality at one-year seems to be lower after EVAS when compared to EVAR. Ongoing, low grade, inflammation could differ between techniques and induce cardiac damage.

This study is designed to establish whether EVAS results in a reduced post-operative inflammatory response during the first year after surgery, compared to EVAR as assessed by trends in circulating inflammatory cytokine concentration.

Study design: International prospective, comparative, explorative study. Study population: Patients scheduled to undergo infra-renal EVAR with a polyester endograft or EVAS for an infrarenal aortic aneurysm. This is an explorative study and therefore only patients who would normally receive a suitable device as part of standard treatment at the participating institutes will be recruited. Blood samples will be taken at specified time points before and after surgery.

Main study parameters/endpoints: The difference in early post-operative and long term inflammatory response between EVAS and EVAR, measured by the incidence of the post-implant syndrome. To investigate the incidence of the post-implant syndrome, the rise in CRP, WBC and circulating cytokines, at specified time points up to 12 months after surgery and the change in aortic thrombus volume and its relationship with the inflammatory response, measured by cytokines' concentrations.

DETAILED DESCRIPTION:
Endovascular sealing of abdominal aortic aneurysms (EVAS) is a new technique to treat infrarenal abdominal aortic aneurysms (AAA), which can be performed more expeditiously than endovascular aneurysm repair (EVAR). The difference with EVAR is that fixation and seal are provided from polymer filled endobags that are placed in the aneurysmal sac. The post-implantation syndrome (PIS) is the clinical and biochemical expression of an inflammatory response following endovascular repair of an aortic aneurysm. More specifically, the presence of fever (body temperature >38 C for ≥1 day) and leukocytosis (white blood cell count (WBC) >12.000/mL) with negative blood cultures and is occurring in over 30% cases after EVAR. It is related to prolonged hospital stay and elevated CRP levels, that in turn increase the risk on major adverse cardiac events. The literature showed that the magnitude of the post-operative inflammatory response depends on the type of endoprothesis used for EVAR and that EVAS is related to a lower post-operative CRP level, lower white blood counts, a lower temperature and less cardiac complications compared to standard EVAR.

The current study was designed to explore the occurence of the post-implant syndrome after EVAR and EVAS. This study was also designed to unravel the cytokines which are involved in the post-implant syndrome after EVAR and EVAS.

In this international, prospective, explorative study 60 patients who are scheduled for EVAR and 60 patients who are scheduled for EVAS will be included. Blood samples (for WBC and circulating cytokines (TNF-α, Interleukin (IL)-1, 1RA, 6, 10, 18, CRP), Troponin T, HsTnT, NT-pro-BNP)) will be taken at:

* Before induction of anesthesia
* At wound closure
* 24 hours after surgery
* 48 hours after surgery
* 1 month after surgery
* 6 months after surgery
* 12 months after surgery

Patients are finished with the study after 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Elective EVAR/EVAS
* Ability and willingness to provide written informed consent
* Age >50 years

Exclusion Criteria:

* Complex EVAR or EVAS, including iliac branched and supra-renal repairs (pre-planned visceral chimneys, fenestrations or branches)
* Ruptured or symptomatic AAA
* Planned internal iliac artery embolization
* Acute or chronic inflammatory illness (i.e. upper respiratory tract infection)
* Active rheumatoid arthritis
* Inflammatory bowel disease, etc.)
* Inflammatory and mycotic aneurysms
* Planned associated surgical procedure (i.e. iliac conduit, femoral endarterectomy, etc.)
* Previous aortic surgery (open or endovascular)
* Untreated malignancy
* Major surgery six weeks before EVAR/EVAS
* Ongoing or recent immunosuppressive treatment, including corticosteroid use

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory response between EVAS and EVAR | Up to 12 months after surgery.
  The change in early post-operative inflammatory response between EVAS and EVAR, measured by the incidence of the post-implant syndrome.
Change in inflammatory response between EVAS and EVAR | Up to 12 months after surgery.
  The change in long term inflammatory response between EVAS and EVAR, measured by the incidence of the post-implant syndrome.

SECONDARY OUTCOMES:
Change in aortic thrombus volume | Up to 12 months after surgery.
  The change in aortic thrombus volume and its relationship with the inflammatory response, measured by cytokines' concentrations.
Pyrexia post operative | 24 to 48 hours after surgery
  Post-operative pyrexia, measured at 24 and 48 hours.
30-day Morbidity | Up to 30 days after surgery
  30-day morbidity measured by cytokines' concentrations.
1 year morbidity | Up to 12 months after surgery.
  1 year morbidity measured by cytokines' concentrations.
Cardiac complications | Up to 12 months after surgery.
  Cardiac complications (including measures of Troponin T, hsTnT, NT-proBNP) measured by cytokines' concentrations.
Mortality | Up to 12 months after surgery.
  (all-cause and cardiac) mortality measured by cytokines' concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, Principal Investigator — Rijnstate Hospital
Locations (7):
- Marienhospital Kevelaer, Kevelaer, Germany
- Rijnstate, Arnhem, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Poland (3):
  - University Hospital No.1, Bydgoszcz
  - Szpital Wojewódzki nr 4, Bytom
  - Institution Hematologii I Transfuzjologii,, Warsaw
- Hospital Universitari I Politècnic La Fe, Valencia, Spain